CLINICAL TRIAL: NCT06840990
Title: Ophthalmic Solution in Corneal Re-epithelization
Brief Title: Cross-linked CMC and Silk Proteins in Corneal Re-epithelization
Acronym: CLCS
Status: Completed | Type: Observational
Sponsor: D&V FARMA srl (Industry)
Collaborators: San Giovanni Addolorata Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: COR-WH
Record Dates: First submitted 2025-02-18; First posted 2025-02-21 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-09

CONDITIONS: Corneal Epithelial Wound Healing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CXC-SP: subjects who underwent either PRK, CXL, PTK or experienced a corneal abrasion treated with a standard therapy plus silk protein and CX-CMC-based eye drops.
  Interventions: Device: CXC-SP
- CTRL: subjects who underwent either PRK , CXL , PTK , or experienced a corneal abrasion. The subjects were treated with the standard therapy only.
  Interventions: Device: CTRL

INTERVENTIONS:
Device: CXC-SP — Standard therapy plus sterile Isotonic ophthalmic solution based on CX-CMC and silk protein, istilled six time a day until complete healing.
  Groups: CXC-SP
Device: CTRL — Standard therapy plus sterile ophtalmic isotonic solution for six time a day until complete healing.
  Groups: CTRL

SUMMARY:
Data analyses and revision of the corneal re-epithelization in patients who underwent either PRK (Photorefractive Keratectomy), CXL (Corneal Cross-Linking), PTK (phototherapeutic keratectomy), or experienced a corneal abrasion. A novel ophthalmic solution containing cross-linked CMC (CX-CMC) and Silk Proteins (SP) has been made available on the market. Both molecules have been widely studied for their wound healing properties in the ophtalmic field. This new ophthalmic solution is the first on the market formulated with a CX-CMC and SP.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had undergone surgical procedures involving de-epithelialization, which included CXL, PRK, and PTK, as well as those with a first diagnosis of corneal abrasion

Exclusion Criteria:

* patients with known allergies or hypersensitivity to any components of the tested formulations or standard therapies, or those requiring different treatments compared to the rest of the study population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data derived from subject who undergone surgical procedures involving de-epithelialization, which included CXL, PRK, and PTK, as well as those with a first diagnosis of corneal abrasionand treated with the ophthalmic solution containing CX-CMC and SP and with lubricant eye drops will be collected and analysed.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Corneal re-ephitalization | 2 WEEKS
  To evaluate and follow the corneal re-ephitalization process a topograph measuring epithelium thickness will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- San Giovanni-Addolorata Hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdel-Naby W, Cole B, Liu A, Liu J, Wan P, Schreiner R, Infanger DW, Paulson NB, Lawrence BD, Rosenblatt MI. Treatment with solubilized Silk-Derived Protein (SDP) enhances rabbit corneal epithelial wound healing. PLoS One. 2017 Nov 20;12(11):e0188154. doi: 10.1371/journal.pone.0188154. eCollection 2017. PMID 29155856
- [Background] Garrett Q, Simmons PA, Xu S, Vehige J, Zhao Z, Ehrmann K, Willcox M. Carboxymethylcellulose binds to human corneal epithelial cells and is a modulator of corneal epithelial wound healing. Invest Ophthalmol Vis Sci. 2007 Apr;48(4):1559-67. doi: 10.1167/iovs.06-0848. PMID 17389485
- [Background] Kundu J, Mohapatra R, Kundu SC. Silk fibroin/sodium carboxymethylcellulose blended films for biotechnological applications. J Biomater Sci Polym Ed. 2011;22(4-6):519-39. doi: 10.1163/092050610X487864. Epub 2010 Jun 21. PMID 20566044
- [Background] Tran SH, Wilson CG, Seib FP. A Review of the Emerging Role of Silk for the Treatment of the Eye. Pharm Res. 2018 Nov 5;35(12):248. doi: 10.1007/s11095-018-2534-y. PMID 30397820
- [Background] Lee JS, Lee SU, Che CY, Lee JE. Comparison of cytotoxicity and wound healing effect of carboxymethylcellulose and hyaluronic acid on human corneal epithelial cells. Int J Ophthalmol. 2015 Apr 18;8(2):215-21. doi: 10.3980/j.issn.2222-3959.2015.02.01. eCollection 2015. PMID 25938030